CLINICAL TRIAL: NCT02829853
Title: Clinical and Genetic Study of Familial Sarcoidosis (SARCFAM)
Acronym: SARCFAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: D50604
Record Dates: First submitted 2016-07-04; First posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Sarcoidosis
Keywords: SARCOIDOSIS; GRANULOMA DISEASES; GENETICS; PREDISPOSITION; EXOME (WES-NGS)
MeSH Terms: conditions — Sarcoidosis; Disease Susceptibility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For main index cases in familial forms of sarcoidosis, two 1 ml samples of frozen PBMC (peripheral blood mononuclear cells) have been included in the bio bank of the diagnosis laboratory (Molecular genetics - GH-HEH - LYON - F)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- sporadic cases (SP): Sporadic cases are defined as patients diagnosed for sarcoidosis, for which the familial history did not reveal any other cases, whatever the relative degree is: 1, 2, 3 or 4. The clinical follow-up and the genetic studies performed in the frame of this project are the same as for the familial group. During the regular follow-up, patients are regularly questioned about the putative occurrence of the disease in their family, and if such a situation occurred, the patient (and his relative) may change from the SP to the familial (FAM) group. In blood samples, genetic analysis by SANGER and WHOLE EXOME NEXT GENERATION SEQUENCING will be done.
  Interventions: Genetic: Genetic analysis by SANGER and WHOLE EXOME NEXT GENERATION SEQUENCING
- familial cases (FAM): Familial cases are defined as patients diagnosed for sarcoidosis with a first and/or second degree relative parent also affected by a well-proven sarcoidosis syndrome. More than 70% of SARCFAM families included two first-degree affected individuals, with both a vertical or horizontal transmission. The Mendelian trait seems to be autosomal dominant. 20 to 30% of the families consists of 3, 4 or more cases, with a subset of families including more than 5 cases. Patients are managed as for the sporadic one, and in such families, an informed consent was also provided with a clear explanation on the complexity of the genetic background of the disease. In blood samples, genetic analysis by SANGER and WHOLE EXOME NEXT GENERATION SEQUENCING will be done.
  Interventions: Genetic: Genetic analysis by SANGER and WHOLE EXOME NEXT GENERATION SEQUENCING

INTERVENTIONS:
Genetic: Genetic analysis by SANGER and WHOLE EXOME NEXT GENERATION SEQUENCING — Patients with sarcoidosis patients are monitored in the regular follow-up in one of 28 GSF clinical centers. Blood sampling was performed in two 5ml classical heparinized tube, as used for red/white/platelets blood cells analysis. The patients receive complete information on the SARCFAM protocol and sign an informed consent stating that the genetic study will be conducted on the BTNL2 gene and genes related to immunity, including loci other than BTNL2.DNA was extracted from a 1-5 ml sample of blood and stored in frozen conditions until analysis. Genomic DNA is captured using Agilent in-solution enrichment methodology (Human Clinical Research Exome, Agilent) with their biotinylated oligonucleotides probes library, followed by paired-end 75 bases massively parallel sequencing on Illumina HiSEQ 400. For each genomic position, the exomic frequencies (Homo & HTZ) are determined from all the exomes already sequenced and/or the exome results provided by 1000G, EVS, HapMap database.

SUMMARY:
Major impacts of air pollution are lung diseases such as granulomatous diseases and mainly sarcoidosis. Understanding the respective role of inorganic / nanoparticles and genetic background in these chronic diseases is a major challenge for the management of patients and prevention strategies. Granulomas are characterized by giant epithelioid and multinucleated cells, reflecting a severe disturbance in immunological pathways induced both by toxic exposure and genetic predisposition. Previous studies demonstrated that professional environmental context and acute exposures (the World Trade Center disaster) to micro/nanoparticles have a pathogenic impact with a sharp increase in sarcoidosis. Sarcoidosis is a multifactorial disease occurring in a genetically vulnerable context. Many gene variants have been linked to an increased odds-ratio of the disease, such BTNL2, CCDC88B, ANNEXIN A11 involved in regulation of T-cell activation and maturation pathways. We have contributed since 2008 to a national cohort (GSF, 28 centers) of ≈ 800 sarcoidosis patients with familial and sporadic presentation of the disease. This collection has been an exceptional (and worldwide unique) tool for the implementation of an exhaustive clinical database on sarcoidosis, modelling of disease evolution and identification of clinical / genetic criteria differentiating sporadic and familial forms.

The main goals of the project are:

1. Completion of the genetic data in order to establish a pattern of gene variants segregating with familial forms of the disease, compared to sporadic one. This will be done by WES (WHOLE EXOME) analysis on the previously collected DNA samples. The informed consent for the patients included the information about the BTNL2 gene, which has been already tested since 2008, and related genes connected to immune pathways, thus allowing a unambiguous information about the research finality of the project.
2. Completion of the clinical data about each patient, in cooperation with the GSF network, management of the database established since 2008. The data collected are those which are commonly detailed in the normal follow-up of the patients. The project do not include any new interventions on the patient (neither radiological or invasive tests).
3. Specific biological studies might be done on the white blood cells of the patients, and might need in such cases a new blood sampling, both in patients and first degree related healthy controls. Theses specific studies will be presented to an ethical committee (CCP) in order to validate the feasibility in term of 'new intervention' on the cohort. The samples collected will be at the same volume of a classical blood sampling (2*7 ml).
4. Any other projects, submitted to the GSF network will needed a specific registration and ethical committee validation.

ELIGIBILITY:
Inclusion Criteria:

* patient affected by sarcoidosis, as defined by clinical criteria such as : chest X-ray staging, pulmonary function tests, biological variables: serum calcium and creatinine, bronchial alveolar lavage cell count and when available, an histological confirmation of the granuloma by biopsy. The disease may be expressed initially as uveitis, cutaneous or other anatomical sites involvement, which must be also confirmed as sarcoidosis-related granuloma by competent pathologists.

Exclusion Criteria:

* Any other disease suggesting sarcoidosis and expressed by similar symptoms, as for ex. hilar lymphadenopathy, other forms of uveitis, restrictive pulmonary syndromes .. etc ….
* Any patients for which the follow-up was not available over the 8 year program of the GSF SARCFAM
* age < 8 years old or > 80 years old

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient affected by sarcoidosis
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2008-01; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
number of mutations founded in the IL34-TIAM gene | Day 0
  Determination of the number of mutations founded in the IL34-TIAM gene which has been described as involved in the formation of granuloma, a key lesion of sarcoidosis

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon / Hopital Edouard Herriot, Lyon, France

REFERENCES:
- [Derived] Calender A, Rollat Farnier PA, Buisson A, Pinson S, Bentaher A, Lebecque S, Corvol H, Abou Taam R, Houdouin V, Bardel C, Roy P, Devouassoux G, Cottin V, Seve P, Bernaudin JF, Lim CX, Weichhart T, Valeyre D, Pacheco Y, Clement A, Nathan N; in the frame of GSF (Groupe Sarcoidose France). Whole exome sequencing in three families segregating a pediatric case of sarcoidosis. BMC Med Genomics. 2018 Mar 6;11(1):23. doi: 10.1186/s12920-018-0338-x. PMID 29510755